CLINICAL TRIAL: NCT01290419
Title: A Phase 1 Randomized, Observer-Blinded,Placebo-Controlled Trial to Evaluate the Safety and Immunogenicity of a Recombinant Respiratory Syncytial Virus F Protein Particle Vaccine in Healthy Adults
Brief Title: Safety Study of Respiratory Syncytial Virus (RSV)-Fusion (F) Protein Particle Vaccine
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Novavax (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: NVX 757.101
Record Dates: First submitted 2011-02-02; First posted 2011-02-07 (Estimated); Last update posted 2012-03-08 (Estimated); Status verified 2012-03

CONDITIONS: Respiratory Syncytial Virus Infections
Keywords: RSV
MeSH Terms: conditions — Respiratory Syncytial Virus Infections

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (7):
- A: Dose 1 + adjuvant (Experimental)
  Interventions: Biological: RSV-F Particle Vaccine
- B: Dose 2 + adjuvant (Experimental)
  Interventions: Biological: RSV-F Particle Vaccine
- C: Dose 3 + adjuvant (Experimental)
  Interventions: Biological: RSV-F Particle Vaccine
- D: Dose 3 alone (Experimental)
  Interventions: Biological: RSV-F Particle Vaccine
- E: Placebo control (Placebo Comparator)
  Interventions: Biological: Placebo
- F: Dose 4 alone (Experimental)
  Interventions: Biological: RSV-F Particle Vaccine
- G: Dose 4 +adjuvant (Experimental)
  Interventions: Biological: RSV-F Particle Vaccine

INTERVENTIONS:
Biological: RSV-F Particle Vaccine — Dose 1 + adjuvant / dose; Day 0 and Day 30
  Arms: A: Dose 1 + adjuvant
Biological: RSV-F Particle Vaccine — Dose 2 + adjuvant / dose; Day 0 and Day 30
  Arms: B: Dose 2 + adjuvant
Biological: RSV-F Particle Vaccine — Dose 3 + adjuvant / dose; Day 0 and Day 30
  Arms: C: Dose 3 + adjuvant
Biological: RSV-F Particle Vaccine — Dose 3 / dose; Day 0 and Day 30
  Arms: D: Dose 3 alone
Biological: Placebo — Placebo; Day 0 and Day 30
  Arms: E: Placebo control
Biological: RSV-F Particle Vaccine — Dose 4 / dose; Day 0 and Day 30
  Arms: F: Dose 4 alone
Biological: RSV-F Particle Vaccine — Dose 4 + adjuvant / dose; Day 0 and Day 30
  Arms: G: Dose 4 +adjuvant

SUMMARY:
A Phase 1, Randomized, Placebo-Controlled, Observer-Blinded, Escalating Dose-Ranging Study to Assess the Safety, and immunogenicity of 6 different recombinant RSV-F formulations in healthy adults (18 to 49 years of age).

Study Objectives:

Primary:

* To assess and compare the safety, reactogenicity, and tolerability of 6 RSV-F protein particle vaccine formulations.

Secondary:

* To assess and compare the immunogenicity (neutralizing antibody and total anti-F antibody) of the 6 RSV-F protein particle vaccine formulations
* To confirm the "dose sparing" and "value added" effects of the aluminum phosphate adjuvant

DETAILED DESCRIPTION:
A total of 150 subjects will be allocated to 7 cohorts. Subjects will be randomly assigned to vaccine treatment or saline placebo in a 4:1 ratio, such that each cohort will include 20 subjects who receive active vaccine (Groups A, B, C, D, F and G) and 5 subjects who receive placebo (Group E).

Subjects will be followed for all AEs, including SAEs and non-serious AEs, from the time of each vaccination through 30 days following the second vaccination (Day 60±5). After Day 60, subjects will be contacted via telephone on a monthly basis (approximately Days 90, 120, 150, 180, and 210) and asked about the occurrence of SAEs and SNMCs.

ELIGIBILITY:
Inclusion Criteria:

* Male or female aged 18 to 49 years inclusive
* Ability to provide written informed consent to participate
* Healthy, as determined by medical history, physical examination, vital signs, and clinical safety laboratory examinations at baseline
* Females are required to fulfill one of the following criteria:

  * At least 1 year post-menopausal
  * Surgically sterile
  * Willing to use oral, implantable, transdermal or injectable contraceptives for 30 days prior to first vaccination and until 28 days after each vaccination
  * Willing to abstain from sexual intercourse or use another reliable form of contraception approved by the Investigator (eg, intrauterine device, female condom, and diaphragm with spermicide, cervical cap, use of condom by the sexual partner, or a sterile sexual partner) for study duration and until 28 days after vaccination
* All female subjects must have a negative urine pregnancy test within 48 hours preceding receipt of each vaccination.
* Comprehension of the study requirements, expressed availability for the required study period, and ability to attend scheduled visits and be contacted by telephone throughout the follow-up period

Exclusion Criteria:

* Presence of significant uncontrolled medical or psychiatric illness (acute or chronic). This includes institution of new medical or surgical treatment, or a significant dose alteration for uncontrolled symptoms or drug toxicity within 3 months of screening and reconfirmed on Day 1 prior to vaccination
* Positive serology for HIV-1 or HIV-2, or HBsAg or HCV antibodies
* Pregnant or lactating female
* Females who plan to become pregnant or plan to discontinue contraceptive precautions within 30 days prior to first vaccination and 28 days after each vaccination
* Cancer, or treatment for cancer, within 3 years, excluding basal cell carcinoma or squamous cell carcinoma, which is allowed
* Presence of any medical condition that may be associated with impaired immune responsiveness, including diabetes mellitus
* Receipt (or history of receipt), during the preceding 3-month period, of any medications or other treatments that may adversely affect the immune system such as allergy injections, immune globulin, interferon, immunomodulators, cytotoxic drugs or other drugs known to be frequently associated with significant major organ toxicity, or systemic corticosteroids (oral or injectable). Inhaled and topical corticosteroids will be allowed.
* Receipt or planned administration of a nonstudy vaccine within 30 days prior to vaccination or during the study. If a nonstudy vaccine has been administered, administration of study vaccine injection can be delayed and given as soon as allowable within the 30-day window, provided the nonstudy vaccine is not administered within 2 weeks prior to study enrollment. Immunization with Tetanus Toxoids Adsorbed for adult use (Td or Tdap) vaccine, on an emergency basis, up to 8 days before or at least 8 days after a dose of study vaccine will be allowed.
* History of illicit drug or alcohol abuse within the previous 1 year or positive drug or alcohol screen
* History of anaphylactic type reaction to injected vaccines
* Receipt of any investigational product or nonregistered drug within the 30 days prior to vaccination or current enrollment in any investigational drug study or intent to enroll in such a study within the ensuing study period
* Receipt or donation of blood or blood products 8 weeks prior to vaccination or planned receipt or donation during the study period
* Acute disease, defined as the presence of a moderate or severe illness (as determined by the Investigator through medical history and physical examination) with or without fever, or an oral temperature of ≥38ºC, within 72 hours prior to vaccination. Study vaccine can be administered to persons with a minor illness, such as diarrhea or mild upper respiratory tract infection with or without low-grade fever. Vaccination can be delayed until the subject has recovered.
* Any condition that, in the opinion of the Investigator, would interfere with the primary study objectives

Ages: 18 Years to 49 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 150 (Actual)
Dates: Start 2010-12; Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
To assess and compare the safety, reactogenicity, and tolerability of 6 RSV-F protein particle vaccine formulations. | Day 60 (2 months)
  This primary outcome will be evaluated through an assessment of the following parameters:
  * Immediate AEs
  * Solicited AEs
  * All SAEs and SNMCs
  * Vital signs
  * Laboratory Assessments

SECONDARY OUTCOMES:
To assess and compare the immunogenicity (neutralizing antibody and total anti-F antibody) of the 6 RSV-F protein particle vaccine formulations | Day 60 (2 months)
  This secondary outcome will be assessed in the following manner:
  * Neutralizing antibody against RSV measured in a PRNT assay
  * Total anti-F IgG measured by ELISA by ELISA

CONTACTS AND LOCATIONS:
Overall Officials: D. Nigel Thomas, Ph.D., Study Director — Novavax, Inc.; Dennis Ruff, MD, Principal Investigator — Healthcare Discoveries d/b/a ICON Development Solutions
Locations (1):
- Healthcare Discoveries d/b/a ICON Development Solutions, San Antonio, Texas, United States

REFERENCES:
- [Background] Calder LJ, Gonzalez-Reyes L, Garcia-Barreno B, Wharton SA, Skehel JJ, Wiley DC, Melero JA. Electron microscopy of the human respiratory syncytial virus fusion protein and complexes that it forms with monoclonal antibodies. Virology. 2000 May 25;271(1):122-31. doi: 10.1006/viro.2000.0279. PMID 10814577
- [Background] Collins PL, Mottet G. Post-translational processing and oligomerization of the fusion glycoprotein of human respiratory syncytial virus. J Gen Virol. 1991 Dec;72 ( Pt 12):3095-101. doi: 10.1099/0022-1317-72-12-3095. PMID 1765771
- [Background] Johnson S, Oliver C, Prince GA, Hemming VG, Pfarr DS, Wang SC, Dormitzer M, O'Grady J, Koenig S, Tamura JK, Woods R, Bansal G, Couchenour D, Tsao E, Hall WC, Young JF. Development of a humanized monoclonal antibody (MEDI-493) with potent in vitro and in vivo activity against respiratory syncytial virus. J Infect Dis. 1997 Nov;176(5):1215-24. doi: 10.1086/514115. PMID 9359721
- [Background] Lopez JA, Bustos R, Orvell C, Berois M, Arbiza J, Garcia-Barreno B, Melero JA. Antigenic structure of human respiratory syncytial virus fusion glycoprotein. J Virol. 1998 Aug;72(8):6922-8. doi: 10.1128/JVI.72.8.6922-6928.1998. PMID 9658147
- [Background] Melero JA, Garcia-Barreno B, Martinez I, Pringle CR, Cane PA. Antigenic structure, evolution and immunobiology of human respiratory syncytial virus attachment (G) protein. J Gen Virol. 1997 Oct;78 ( Pt 10):2411-8. doi: 10.1099/0022-1317-78-10-2411. No abstract available. PMID 9349459
- [Background] Thompson WW, Shay DK, Weintraub E, Brammer L, Cox N, Anderson LJ, Fukuda K. Mortality associated with influenza and respiratory syncytial virus in the United States. JAMA. 2003 Jan 8;289(2):179-86. doi: 10.1001/jama.289.2.179. PMID 12517228
- [Background] U.S. Department of Health and Human Services, Food and Drug Administration, Center for Biologics Evaluation and Research. Toxicity Grading Scale for Healthy Adult and Adolescent Volunteers Enrolled in Preventive Vaccine Clinical Trials. September 2007.
- [Derived] Glenn GM, Smith G, Fries L, Raghunandan R, Lu H, Zhou B, Thomas DN, Hickman SP, Kpamegan E, Boddapati S, Piedra PA. Safety and immunogenicity of a Sf9 insect cell-derived respiratory syncytial virus fusion protein nanoparticle vaccine. Vaccine. 2013 Jan 7;31(3):524-32. doi: 10.1016/j.vaccine.2012.11.009. Epub 2012 Nov 12. PMID 23153449